CLINICAL TRIAL: NCT04154007
Title: Acute Kidney Injury in Patients With Acute Respiratory Distress Syndrome: Incidence, Risk Factors and Its Impact on the Outcome
Brief Title: Acute Kidney Injury in Patients With Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, Lecturer of anesthesia and surgical intensive care, Zagazig University
Other Study IDs: 5670/17-10-2019
Record Dates: First submitted 2019-11-03; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Acute Kidney Injury; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Acute Kidney Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Patients who met the diagnosis of ARDS: ARDS patients were followed for the development of AKI during their ICU stay
  Interventions: Diagnostic Test: kidney function tests - urine output

INTERVENTIONS:
Diagnostic Test: kidney function tests - urine output — AKI was classified based on the worst of either creatinine or urine output criterion as follows:
  Stage I 1.5-1.9 times baseline OR ≥0.3 mg/dl increase in the serum creatinine, OR urine output <0.5 ml/kg per hour for 6 to 12 hours.
  Stage II 2.0-2.9 times baseline increase in the serum creatinine OR urine output <0.5 ml/kg per hour for ≥12 hours.
  Stage III 3.0 times baseline increase in the serum creatinine OR increase in serum creatinine to ≥4.0 mg OR urine output of <0.3 ml/kg per hour for ≥24 hours, OR anuria for ≥12 hours OR the initiation of renal replacement therapy.

SUMMARY:
Several studies suggested that ARDS may have important adverse effects on renal function, but few studies have specifically addressed the risk factors of AKI and its impact on the outcome in theses patients.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome is considered an acute diffuse lung injury in which an inciting inflammatory event is followed by hypoxemic respiratory failure. Despite advances in the management of ARDS, the mortality remains high. The LUNG SAFE study reported that hospital mortality was 34.9% in patients with mild ARDS, 40.3% in patients with moderate ARDS, and 46.1% in patients with severe ARDS. Understanding the prognostic factors in ARDS is essential for decreasing its mortality. Acute kidney injury (AKI) is a common and challenging medical condition in critically ill patients, in which there is a sudden renal impairment during hours to days and it is known to be associated with increased mortality .Other adverse outcomes associated with AKI includes chronic kidney disease (CKD) and high cardio-vascular complications. The incidence of AKI in hospitalized adults was reported to be 22% with a mortality rate of 24%. The severity of AKI ranges from stage 1 to stage 3 according to The KDIGO (Kidney Disease: Improving Global Outcomes) system, based on decreased urine output over time, or increases in serum creatinine, or both.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients (≥18 years old)
* diagnosis of ARDS according to Berlin definition

Exclusion Criteria:

* Patients with preexisting chronic kidney disease
* AKI prior to the onset of ARDS

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 81 ARDS patients admitted to the Respiratory, Surgical and Internal Medicine Intensive Care unit, Zagazig University Hospitals during the period from September 2017 to March 2019
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
development of AKI | 30 days
  AKI was classified based on the worst of either creatinine or urine output criterion as follows:
  Stage I 1.5-1.9 times baseline OR ≥0.3 mg/dl increase in the serum creatinine, OR urine output <0.5 ml/kg per hour for 6 to 12 hours.
  Stage II 2.0-2.9 times baseline increase in the serum creatinine OR urine output <0.5 ml/kg per hour for ≥12 hours.
  Stage III 3.0 times baseline increase in the serum creatinine OR increase in serum creatinine to ≥4.0 mg OR urine output of <0.3 ml/kg per hour for ≥24 hours, OR anuria for ≥12 hours OR the initiation of renal replacement therapy.

SECONDARY OUTCOMES:
ICU length of stay. | 30 days
  development of AKI affects the ICU stay
hospital length of stay. | 90 days
  development of AKI may affect the length of stay in hospital
Hospital mortality | 90 days
  the effect of development of AKI on the mortality of ARDS patients

CONTACTS AND LOCATIONS:
Overall Officials: Eman Shebl, MD, Study Director — Chest department, Faculty of Medicine, Zagazig University; Lamiaa G Zake, MD, Principal Investigator — Chest department, Faculty of Medicine, Zagazig University; Sherif MS Mowafy, MD, Principal Investigator — Anesthesia and Surgical Intensive Care department, Faculty of Medicine, Zagazig University; Ayman R Abd El-Hameed, MD, Principal Investigator — Nephrology Internal Medicine department, Faculty of Medicine, Zagazig University
Locations (1):
- Respiratory, Surgical, Internal medicine ICUs, Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available within 6 months after publication
Access Criteria: by contacting the study director

REFERENCES:
- [Background] Peter JV, John P, Graham PL, Moran JL, George IA, Bersten A. Corticosteroids in the prevention and treatment of acute respiratory distress syndrome (ARDS) in adults: meta-analysis. BMJ. 2008 May 3;336(7651):1006-9. doi: 10.1136/bmj.39537.939039.BE. Epub 2008 Apr 23. PMID 18434379
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Cartin-Ceba R, Haugen EN, Iscimen R, Trillo-Alvarez C, Juncos L, Gajic O. Evaluation of "Loss" and "End stage renal disease" after acute kidney injury defined by the Risk, Injury, Failure, Loss and ESRD classification in critically ill patients. Intensive Care Med. 2009 Dec;35(12):2087-95. doi: 10.1007/s00134-009-1635-9. Epub 2009 Sep 15. PMID 19756503
- [Background] Hoste EA, Schurgers M. Epidemiology of acute kidney injury: how big is the problem? Crit Care Med. 2008 Apr;36(4 Suppl):S146-51. doi: 10.1097/CCM.0b013e318168c590. PMID 18382186
- [Background] Coca SG, Cho KC, Hsu CY. Acute kidney injury in the elderly: predisposition to chronic kidney disease and vice versa. Nephron Clin Pract. 2011;119 Suppl 1(Suppl 1):c19-24. doi: 10.1159/000328023. Epub 2011 Aug 10. PMID 21832852
- [Background] Susantitaphong P, Cruz DN, Cerda J, Abulfaraj M, Alqahtani F, Koulouridis I, Jaber BL; Acute Kidney Injury Advisory Group of the American Society of Nephrology. World incidence of AKI: a meta-analysis. Clin J Am Soc Nephrol. 2013 Sep;8(9):1482-93. doi: 10.2215/CJN.00710113. Epub 2013 Jun 6. PMID 23744003
- [Background] Fischer MJ, Brimhall BB, Lezotte DC, Glazner JE, Parikh CR. Uncomplicated acute renal failure and hospital resource utilization: a retrospective multicenter analysis. Am J Kidney Dis. 2005 Dec;46(6):1049-57. doi: 10.1053/j.ajkd.2005.09.006. PMID 16310570
- [Background] Kidney Disease: Improving global outcomes (KDIGO) acute kidney injury working group. KDIGO clinical practice guideline for acute kidney injury. Kidney Int Suppl (2012). 2012;2(1):1-138.
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Hoste EA, Clermont G, Kersten A, Venkataraman R, Angus DC, De Bacquer D, Kellum JA. RIFLE criteria for acute kidney injury are associated with hospital mortality in critically ill patients: a cohort analysis. Crit Care. 2006;10(3):R73. doi: 10.1186/cc4915. Epub 2006 May 12. PMID 16696865